CLINICAL TRIAL: NCT00203203
Title: Randomized Controlled Single Blind Trial of Autologous Bone Marrow Mononuclear Cells Under Electromechanical Guidance for Therapeutic Angiogenesis
Brief Title: Autologous Stem Cells for Cardiac Angiogenesis (FOCUS HF)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Texas Heart Institute (Other)
Collaborators: CHI St. Luke's Health, Texas (Other)
Responsible Party: Principal Investigator, Emerson Perin, MD, PhD, Director Clinical Research for Cardiovascular Medicine and Director Stem Cell Center, Texas Heart Institute
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HSC-MS-04-141
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Results first posted 2013-01-30 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-10

CONDITIONS: Ischemic Cardiomyopathy
Keywords: Autologous; Cardiac; Stem Cell; Transplant
MeSH Terms: interventions — Crossing Over, Genetic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stem Cell Therapy (Experimental): Subject is randomized to receive Stem Cell Therapy (intramyocardial injection of stem cells) via NOGA mapping.
  Interventions: Device: Intramyocardial Injection of stem cells via NOGA Mapping
- Control, then Stem Cell Therapy (Other): Subject is randomized to receive a NOGA mapping and no injections at time of active enrollment.
  At 6 months, subject is offered stem cell therapy.
  Interventions: Other: Control, then Stem Cell Therapy

INTERVENTIONS:
Device: Intramyocardial Injection of stem cells via NOGA Mapping — Subject is randomized to receive intramyocardial injection of stem cells (stem cell therapy) via NOGA mapping to deliver cells in the active arm of the protocol.
  Other Names: NOGA Star catheter and Myostar Injection.
  Arms: Stem Cell Therapy
Other: Control, then Stem Cell Therapy — Subject is randomized to receive a NOGA mapping and no injections (sham treatment)at time of active enrollment and treatment then offered stem cell therapy at 6 months.
  Other Names: cross-over
  Arms: Control, then Stem Cell Therapy

SUMMARY:
This is a phase 1, single-blind trial to evaluate using autologous bone marrow mononuclear stem cells in ischemic cardiomyopathy patients. The patients must have a Left Ventricular Ejection Fraction (LVEF) of less than or equal to 45%. Once the patient meets all inclusion criteria, and no exclusion criteria are found, the subject is consented for the study, and extensive baseline testing is performed at St Luke's Hospital in Houston. Once all baseline testing criteria is met, the patient has their own bone marrow harvested and later that day the subject is taken to a cardiac catheterization lab where left ventricular electromechanical mapping using NOGA software (NOGA mapping) is performed and the processed stem cells are injected under electromechanical guidance into the affected areas of the left ventricle. The patient is usually discharged home the next day and returns for follow up visits at weeks 1, 2, 4, 6, 8, 12, months 6 and 12 and for phone call follow-up at months 4, 5, 7, 8, 9, 10, 11. Patients undergo extensive testing at most of these follow-up visits, including repeat cardiac catheterization with NOGA mapping at month 6 after stem cell injection.

DETAILED DESCRIPTION:
This is a phase 1, single-blind trial to evaluate the use of autologous bone marrow mononuclear stem cells in ischemic cardiomyopathy patients. The study hypothesis is that transendocardial injections of autologous mononuclear bone marrow cells in patients with end-stage ischemic heart disease is safe, can promote neovascularization, and can improve perfusion and myocardial contractility. The primary object of this study will be to evaluate the safety of autologous-bone-marrow mononuclear cell injections. The secondary endpoint of the study is to assess the efficacy of autologous bone marrow cells in improving cardiac contractile function and functional outcome. The efficacy will be assessed on the basis of the treadmill Max VO2 (maximum volume oxygen uptake). Secondarily the efficacy will be assessed on the basis of clinical status and imaging rests, with follow-up extending to 1 year after enrollment.A maximum of 30 patients will be enrolled in the study. At the end of the 6-month visit. after the required angiogram with mapping and non-invasive testing is complete, the patients will be told whether they were in the control or the active group (stem cell therapy). Those in the control group will be told before final invasive testing, and those who consent may cross over to the active therapy arm and undergo the cell injection procedure (control, then stem cell therapy. In these patients, the foll-up angiogram and mapping procedure will also serve as the baseline procedure required for cell injection. Bone marrow mononuclear cells will be injected in an identical fashion, according to the same criteria described for the original treatment group, and these patients will have identical follow-up visits starting again at the baseline time-point and extending for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* LVEF less than 45%
* Functional class III or IV angina
* At least 7% reversibility by Single Photon Emission Computed Tomography (SPECT) nuclear study
* there are additional inc. criteria

Exclusion Criteria:

* AGe <18 or >70 years of age
* Constant atrial fibrillation
* Left ventricular (LV) thrombus
* History of malignancy in the last 5 years
* LV wall thickness of < 8 mm at the target site
* there are additional exclusion criteria

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2004-04; Primary Completion 2008-08 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emerson Perin, MD,PhD., Principal Investigator — Texas Heart Institute/Baylor St Luke's Medical Center
Locations (1):
- Texas Heart Institute/Baylor St. Luke's Medical Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Data summarized and published. No need to share individual patient data.

REFERENCES:
- [Result] Perin EC, Silva GV, Henry TD, Cabreira-Hansen MG, Moore WH, Coulter SA, Herlihy JP, Fernandes MR, Cheong BY, Flamm SD, Traverse JH, Zheng Y, Smith D, Shaw S, Westbrook L, Olson R, Patel D, Gahremanpour A, Canales J, Vaughn WK, Willerson JT. A randomized study of transendocardial injection of autologous bone marrow mononuclear cells and cell function analysis in ischemic heart failure (FOCUS-HF). Am Heart J. 2011 Jun;161(6):1078-87.e3. doi: 10.1016/j.ahj.2011.01.028. Epub 2011 May 10. PMID 21641354
- See also: Stem Cell Group at Texas Heart Institute — http://www.texasheart.org/stemcell

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty patients were recruited between 4/14/04 and 2/8/07 from outpatient cardiology clinics.
Groups:
- Stem Cell Therapy: Subject is randomized to receive intramyocardial injection of stem cells (stem cell therapy) via NOGA mapping.
Period: Overall Study
Arm/Group | Control, Then Stem Cell Therapy | Stem Cell Therapy
Started | 10 | 20
Completed | 9 | 20
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control, Then Stem Cell Therapy | Stem Cell Therapy | Total
Number analyzed (Participants) | 10 | 20 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 14 | 24
  >=65 years | 0 | 6 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.3 (8.6) | 60.5 (6.4) | 60.0 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 7 | 15 | 22
Region of Enrollment [Number; unit: participants]
  United States | 10 | 20 | 30

OUTCOME MEASURES:

1. Primary Outcome: Safety of Autologous-bone-marrow Injections
Description: Safety of cell injections was assessed by reviewing adverse events at 3 time points: (1) up to 2 weeks post-procedure), (2) 3 months post-procedure, and (3) at 6 months post-procedure. Major adverse events were adjudicated (hospitalization, arrhythmia, exacerbation of congestive HF [CHF], acute coronary syndrome, myocardial infarction, stroke, or death).
Time Frame: up to 2 weeks post-procedure, 3 months and 6 months
Population: Adverse events which occurred in all participants.
Measure: Number; unit: participants
Arm/Group | Control, Then Stem Cell Therapy | Stem Cell Therapy
Number analyzed (Participants) | 10 | 20
participants
  post-procedural transient left bundle branch block | 1 | 1
  Post-procedure pericardial effusion (nonsignifiant | 0 | 1
  Post-procedure transient fever | 1 | 0
  Fever (6 months) | 2 | 0
  Sustained ventricular arrhythmias (6 months) | 0 | 0
  Discharge implantable cardiac defibrillator (6 mo) | 0 | 1
  Exacerbation of congestive heart failure (6 mo) | 1 | 2
  Myocardial infarction (6 months) | 0 | 0
  Death (6 months) | 0 | 0

2. Secondary Outcome: Canadian Cardiovascular (CCS) Angina Score
Description: Clinical and functional assessment in endstage ischemic cardiomyopathy patients using Canadian Cardiovascular (CCS) Angina Score which indicates discomfort from angina (chest pain).
  Class I- Angina only during strenuous or prolonged activity Class II- Slight limitation, with angina only during vigorous physical activity Class III- Symptoms with everyday living activities (moderate limitation) Class IV- Inability to perform any activity without angina or angina at rest (severe limitation)
Time Frame: baseline, 3 months and 6 months
Population: The data was analyzed for all participants in control and treated groups.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control, Then Stem Cell Therapy | Stem Cell Therapy
Number analyzed (Participants) | 10 | 20
units on a scale
  CCS baseline | 3 (0.3) | 3 (0.2)
  CCS 3 months | 2.2 (0.3) | 2.1 (0.2)
  CCS 6 months | 2.6 (0.3) | 1.8 (0.2)

3. Secondary Outcome: New York Heart Association (NYHA)Classification
Description: Clinical and functional assessment in endstage ischemic cardiomyopathy patients using New York Heart Association (NYHA)Classification and indicates extent of heart failure based on limitations in physical activity.
  Class I- No symptoms/limitation in ordinary physical activity (shortness of breath when walking, etc) Class II-Mild symptoms/slight limitation during ordinary activity Class III- Marked limitation in activity due to symptoms, even during less-than-ordinary activity Class IV- Severe limitations in activity/experiences symptoms while at rest (bedbound)
Time Frame: baseline, 3 months and 6 months
Population: The data was analyzed for all participants in control and treated groups.
Measure: Mean (Standard Deviation); unit: NYHA Functional Class
Arm/Group | Control, Then Stem Cell Therapy | Stem Cell Therapy
Number analyzed (Participants) | 10 | 20
NYHA Functional Class
  NYHA Baseline | 2.6 (0.3) | 2.3 (0.2)
  NYHA 3 months | 1.9 (0.3) | 2 (0.2)
  NYHA 6 months | 2.4 (0.3) | 1.8 (0.2)

4. Secondary Outcome: Myocardial Oxygen Consumption (MVO2)
Description: Clinical and functional assessment in endstage ischemic cardiomyopathy patients using Myocardial Oxygen Consumption (MVO2)which is the amount of oxygen used by the heart muscle and is indicative of heart muscle function. Normal value is 15.5 Volume %. Measured as milliliters (ml) oxygen per kilogram (kg) body weight per minute.
Time Frame: baseline, 3 months and 6 months
Population: The data was analyzed for all participants in control and treated groups.
Measure: Mean (Standard Deviation); unit: Percentage of Oxygen Saturation
Arm/Group | Control, Then Stem Cell Therapy | Stem Cell Therapy
Number analyzed (Participants) | 10 | 20
Percentage of Oxygen Saturation
  MVO2 (ml/kg per min) baseline | 14.8 (0.8) | 14.7 (0.6)
  MVO2 (ml/kg per min) 3 months | 15.7 (0.8) | 15.5 (0.6)
  MVO2 (ml/kg per min) 6 months | 15.6 (0.9) | 15.8 (0.6)

5. Secondary Outcome: Echocardiography (EF)Percent (%)
Description: Clinical and functional assessment in endstage ischemic cardiomyopathy patients using Echocardiography measures ejection fraction(EF)as a percentage(%) of blood leaving the heart with each beat or contraction. It can provide information concerning structural characteristics and blood flow in the heart and blood vessels. A normal heart pumps 50-75% of the blood with each contraction.
Time Frame: baseline, 3 months and 6 months
Population: The data was analyzed for all participants in control and treated groups.
Measure: Mean (Standard Deviation); unit: Ejection Fraction %
Arm/Group | Control, Then Stem Cell Therapy | Stem Cell Therapy
Number analyzed (Participants) | 10 | 20
Ejection Fraction %
  Echocardiography EF (%) baseline | 39 (9.1) | 37 (10.6)
  Echocardiography EF (%) 3 months | 41 (5.4) | 38 (5.4)
  Echocardiography EF (%) 6 months | 42 (5.4) | 40 (5.4)

6. Secondary Outcome: Minute Ventilation- Carbon Dioxide Production Relationship (VE/VCO2 Slope)
Description: Clinical and functional assessment in endstage ischemic cardiomyopathy patients using Minute Ventilation- Carbon Dioxide Production Relationship (VE/VCO2 slope)measure during a cardiopulmonary exercise test has a high prognostic value for survival in heart failure patients. Normal VE (milliliters per minute)/VCO2 (milliliters per minute)equals 25.
Time Frame: baseline and 3 months
Population: The data was analyzed for all participants in control and treated groups.
Measure: Mean (Standard Deviation); unit: VE/VCO2 slope
Arm/Group | Control, Then Stem Cell Therapy | Stem Cell Therapy
Number analyzed (Participants) | 10 | 20
VE/VCO2 slope
  VE/VCO2 baseline | 29.8 (8) | 32.7 (6)
  VE/VCO2 3 months | 32.8 (5) | 31.8 (7)

7. Secondary Outcome: Echocardiography Wall Motion Score Index (WMSI)
Description: Clinical and functional assessment in endstage ischemic cardiomyopathy patients using Echocardiography Wall Motion Score Index (WMSI)which allows detection of abnormalities in the heart wall or blood flowing through the heart. Normal contracting Left Ventricle has WMSI of 1. Larger WMSI indicates higher degree of abnormalities (2 for hypokinetic, 3 for akinetic, 4 for dyskinetic, and 5 for aneurysmal). WMSI was calculated as the sum of scores divided by the total number of segments.
Time Frame: baseline and 3 months
Population: The data was analyzed for all participants in control and treated groups.
Measure: Mean (Standard Deviation); unit: Wall Motion Score Index
Arm/Group | Control, Then Stem Cell Therapy | Stem Cell Therapy
Number analyzed (Participants) | 10 | 20
Wall Motion Score Index
  Wall Motion Score Index (WMSI) baseline | 1.7 (0.5) | 1.7 (0.5)
  Wall Motion Score Index (WMSI) 3 months | 1.6 (0.4) | 1.7 (0.6)

8. Secondary Outcome: Single-photon Emission Computed Tomography (SPECT) Imaging for Left Ventricular Ejection Fraction (LVEF) Percentage (%)
Description: Clinical and functional assessment in endstage ischemic cardiomyopathy patients using Single-photon emission computed tomography (SPECT) imaging for Left Ventricular Ejection Fraction (LVEF) percentage (%)to determine how well the heart is pumping blood from the left ventricle. Different method for evaluating how much (%) of blood is pumped through heart with each contraction.
Time Frame: baseline, 3 months and 6 months
Population: The data was analyzed for all participants in control and treated groups.
Measure: Mean (Standard Deviation); unit: Left Ventricular Ejection Fraction (%)
Arm/Group | Control, Then Stem Cell Therapy | Stem Cell Therapy
Number analyzed (Participants) | 10 | 20
Left Ventricular Ejection Fraction (%)
  SPECT LVEF (%) baseline | 43 (10.4) | 41.5 (11.2)
  SPECT LVEF (%) 3 months | 46.8 (9.5) | 43.2 (11.1)
  SPECT LVEF (%) 6 months | 47.8 (7.5) | 44 (13.4)

9. Secondary Outcome: Angiography Left Ventricular Ejection Fraction (LVEF) Percent (%)
Description: Clinical and functional assessment in endstage ischemic cardiomyopathy patients using angiography left ventricular ejection fraction (LVEF) percent (%) which is an invasive method used to estimate how well the heart is pumping blood through the ventricle and is considered the "gold" standard.
Time Frame: baseline and 6 months
Population: The data was analyzed for all participants in control and treated groups.
Measure: Mean (Standard Deviation); unit: Angiography LVEF (%)
Arm/Group | Control, Then Stem Cell Therapy | Stem Cell Therapy
Number analyzed (Participants) | 10 | 20
Angiography LVEF (%)
  Angiography LVEF (%) baseline | 40 (3.2) | 37.5 (8.2)
  Angiography LVEF (%) 6 months | 40.9 (8.5) | 42 (14.4)

10. Secondary Outcome: Left Ventricular End-Diastolic Volume (LVEDV)
Description: Clinical and functional assessment in endstage ischemic cardiomyopathy patients using Left Ventricular End-Diastolic Volume (LVEDV)which is the volume of blood inside the left ventricle when the heart has completed its filling cycle. The volume of the left ventricle is measured during contraction and relaxation. Normal heart volume inside the left ventricle is about 140 milliliters.
Time Frame: baseline, 3 months and 6 months
Measure: Mean (Standard Deviation); unit: Volume in left ventricle (milliliters)
Arm/Group | Control, Then Stem Cell Therapy | Stem Cell Therapy
Number analyzed (Participants) | 10 | 20
Volume in left ventricle (milliliters)
  LVEDV (ml) baseline | 132.2 (43.6) | 133.2 (53.6)
  LVEDV (ml) 3 months | 125.7 (46.3) | 123.9 (58.2)
  LVEDV (ml) 6 months | 120.0 (30.9) | 123.9 (39.7)

11. Secondary Outcome: Left Ventricular End-Systolic Volume (LVESV) (ml)
Description: Clinical and functional assessment in endstage ischemic cardiomyopathy patients using Left Ventricular End-Systolic Volume (LVESV)when the blood moves from the ventricles to the atria during the contraction cycle. Measured as volume in milliliters (ml). Normal is approximately 60- 65 milliliters.
Time Frame: baseline, 3 months and 6 months
Population: The data was analyzed for all participants in control and treated groups.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Control, Then Stem Cell Therapy | Stem Cell Therapy
Number analyzed (Participants) | 10 | 20
ml
  LVESV (ml) baseline | 81.7 (40.7) | 92.9 (50.5)
  LVESV (ml) 3 months | 74.4 (37) | 83.2 (43.2)
  LVESV (ml) 6 months | 71.8 (27.2) | 74 (29.5)

12. Secondary Outcome: Endocardial Unipolar Voltages (UPV)
Description: Clinical and functional assessment in endstage ischemic cardiomyopathy patients using Endocardial Unipolar Voltages (UPV)in millivolts(mV)which may be indicative of scar tissue. Normal is <5.5 mV.
Time Frame: baseline and 6 months
Population: The data was analyzed for all participants in control and treated groups.
Measure: Mean (Standard Deviation); unit: Unipolar voltage (mV)
Arm/Group | Control, Then Stem Cell Therapy | Stem Cell Therapy
Number analyzed (Participants) | 10 | 20
Unipolar voltage (mV)
  UPV (mV) baseline | 10.2 (4.3) | 10.5 (5.1)
  UPV (mV) 6 months | 10.1 (4.8) | 10.8 (5.4)

13. Secondary Outcome: Linear Local Shortening (LLS)
Description: Clinical and functional assessment in endstage ischemic cardiomyopathy patients using Linear Local Shortening (LLS)which is an indicator of mechanical properties of the heart and measured as a percentage (%)of local contraction.
Time Frame: baseline and 6 months
Measure: Mean (Standard Deviation); unit: percentage of linear local shortening
Arm/Group | Control, Then Stem Cell Therapy | Stem Cell Therapy
Number analyzed (Participants) | 10 | 20
percentage of linear local shortening
  LLS (%) baseline | 12.1 (6.8) | 10.5 (7.3)
  LLS (%) 6 months | 9.1 (6.4) | 10.8 (6.8)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected pre-procedure, during procedure, after procedure, at 1, 2, 4, 6, 8 weeks post procedure and monthly until 1 year post-procedure.
Arm/Group | Control, Then Stem Cell Therapy | Stem Cell Therapy
Serious Adverse Events (participants affected / at risk) | 7/10 | 11/20
Other Adverse Events (participants affected / at risk) | 9/10 | 18/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control, Then Stem Cell Therapy (N=10) | Stem Cell Therapy (N=20)
Chest pain and slightly elevated Troponin I (Cardiac disorders) | 0 (0) | 1 (2)
Confusion/disorientation (Nervous system disorders) | 0 (0) | 1 (1)
Elevated troponin,chestpain and fever with episode of cellulitis (Cardiac disorders) | 0 (0) | 1 (1)
False positive culture on processed stem cells at day 5 (Infections and infestations) | 0 (0) | 1 (1)
Hospitalized for chest pain (Cardiac disorders) | 0 (0) | 1 (1)
Hospitalized for heart failure at one year (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Placement of AICD (Cardiac disorders) | 2 (2) | 1 (1)
Pulmonary edema & slightly elevated Troponin I with ablation of atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Pulmonary edema within 24 hrs of treatment (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Replacement of AICD (Cardiac disorders) | 1 (1) | 2 (2)
Restenosis without symptoms at 6 months, received stent (Cardiac disorders) | 0 (0) | 2 (2)
Staph aureus septicemia (left sternoclavicular area) leg (Infections and infestations) | 1 (1) | 0 (0)
Troponin I elevation in presence of new onset Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Urosepsis (Renal and urinary disorders) | 1 (1) | 0 (0)
back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
bronchitis, decompensated heart failure (Cardiac disorders) | 1 (1) | 0 (0)
decompensated heart failure (Cardiac disorders) | 0 (0) | 1 (1)
elevated Troponin T in presence of bacteremia (Cardiac disorders) | 1 (1) | 0 (0)
supraventricular tachycardia ablation (Cardiac disorders) | 0 (0) | 2 (2)
unstable angina and stent (Cardiac disorders) | 1 (1) | 0 (0)
urosepsis and chest pain (Cardiac disorders) | 1 (1) | 0 (0)
ventricular tachycardia during 6 month F/Ucath requiring cardioversion (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control, Then Stem Cell Therapy (N=10) | Stem Cell Therapy (N=20)
ICD firing (General disorders) | 0 (0) | 1 (1)
abcess left sternovascular joint (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
abcess tooth (Infections and infestations) | 1 (1) | 1 (1)
abdominal bloating (Gastrointestinal disorders) | 1 (1) | 2 (2)
abnormalities/ pain eye (Eye disorders) | 1 (1) | 1 (1)
abnormality on MRI scan (General disorders) | 0 (0) | 1 (1)
albumin, increase (General disorders) | 1 (2) | 0 (0)
anemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
back/ hip pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 9 (16)
bloody nose (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
blurred vision (Eye disorders) | 1 (1) | 0 (0)
bone fracture (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
bone pain, extremities (Musculoskeletal and connective tissue disorders) | 1 (4) | 3 (4)
bronchitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
carbuncles on body (Infections and infestations) | 0 (0) | 1 (1)
carpel tunnel release (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
cellulitis (Infections and infestations) | 0 (0) | 2 (3)
changes in cardiac enzymes (CK-MB,BNP,CRP, troponin) (Cardiac disorders) | 1 (1) | 5 (9)
changes in heart rate (Cardiac disorders) | 2 (3) | 3 (4)
changes in renal enzymes (BUN, creatinine, chloride) (Renal and urinary disorders) | 1 (1) | 2 (2)
chest pain/ increased chest pain (Cardiac disorders) | 4 (6) | 16 (23)
chills (Infections and infestations) | 0 (0) | 1 (1)
chronic obtructive pulmonary disease, increased symptoms (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
cold/ congestion (General disorders) | 2 (2) | 5 (7)
constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (5)
crackles/ wheezes in lungs (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (6)
cramping (Gastrointestinal disorders) | 0 (0) | 1 (1)
decrease in platelets/ hematocrit (Blood and lymphatic system disorders) | 2 (3) | 0 (0)
depression (Psychiatric disorders) | 0 (0) | 1 (1)
diabetes uncontrolled (Endocrine disorders) | 0 (0) | 1 (3)
diaphoresis (General disorders) | 0 (0) | 1 (1)
diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
digestive problems (Gastrointestinal disorders) | 0 (0) | 3 (3)
disorientation (General disorders) | 0 (0) | 1 (1)
dizziness/ light-headedness (General disorders) | 3 (3) | 5 (8)
edema, extremity not specified (Blood and lymphatic system disorders) | 1 (2) | 4 (7)
edema, upper extremities (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
electrocardiogram changes (Cardiac disorders) | 0 (0) | 4 (17)
eyes sensitive to light (Eye disorders) | 1 (1) | 0 (0)
fall/ balance problems (General disorders) | 0 (0) | 3 (3)
fatigue/ weakness (General disorders) | 2 (2) | 7 (11)
fever (General disorders) | 3 (3) | 2 (3)
gastroespohageal reflux (Gastrointestinal disorders) | 0 (0) | 1 (1)
gout, increased symptoms (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
gum bleeding (General disorders) | 1 (1) | 0 (0)
headache (General disorders) | 4 (4) | 4 (4)
heart failure (Cardiac disorders) | 0 (0) | 2 (4)
heart palpitations (Cardiac disorders) | 2 (2) | 2 (2)
heartburn (Gastrointestinal disorders) | 1 (1) | 0 (0)
hematoma at catheter site (General disorders) | 3 (4) | 3 (5)
hyperglycermia (Endocrine disorders) | 1 (1) | 2 (3)
hypertension (Cardiac disorders) | 0 (0) | 6 (6)
hypoglycemia (Endocrine disorders) | 0 (0) | 2 (2)
hypotension (Cardiac disorders) | 0 (0) | 1 (1)
influenza/ flu-like symptoms (Infections and infestations) | 2 (2) | 1 (1)
insomnia/ sleep disorders (General disorders) | 0 (0) | 3 (3)
itching (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
lesion right foot (Infections and infestations) | 1 (1) | 0 (0)
muscle pain/pull (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
myocardial infaction, non-ST elevation (Cardiac disorders) | 0 (0) | 1 (1)
nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
numbness/ tingling in extremities (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (9)
petechia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
pleuritic chest pain (Cardiac disorders) | 0 (0) | 1 (1)
probable obstructive sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
renal insufficiency/ urinary problems (Renal and urinary disorders) | 1 (3) | 0 (0)
sciatica (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
scrotal edema/ erythema (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
shingles (Infections and infestations) | 1 (1) | 0 (0)
shortness of breath, lying down (Cardiac disorders) | 1 (1) | 1 (1)
shortness of breath/ increased shortness of breath/ difficulty breathing (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 7 (9)
shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 4 (4)
sinus congestion/ compliant (General disorders) | 2 (2) | 2 (6)
skin flushing (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
slurred speech/ dysphasia (Nervous system disorders) | 0 (0) | 2 (2)
soreness/ brusing (General disorders) | 0 (0) | 2 (2)
spider bite (General disorders) | 0 (0) | 1 (1)
swelling/ edema lower extremities (Blood and lymphatic system disorders) | 2 (2) | 10 (17)
swelling/ edema upper extremity (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
tremors (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
upper respiratory infection (Infections and infestations) | 0 (0) | 3 (3)
urinary tract infection (Renal and urinary disorders) | 1 (1) | 1 (2)
urinary/ bladder problems (Renal and urinary disorders) | 1 (1) | 1 (2)
virus (Infections and infestations) | 1 (1) | 1 (1)
weight gain (General disorders) | 0 (0) | 3 (3)
white blood count, elevated (Infections and infestations) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The study is a preliminary study based on a small sample size which limits the statistical rigor of the analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No